CLINICAL TRIAL: NCT05848609
Title: Prospective Evaluation of Functional Status and Quality of Life in Older Patients With Colorectal Cancer Undergoing Robotic Surgery
Brief Title: Functional Status and Quality of Life in Older Patients Undergoing Robotic Surgery for Colorectal Cancer
Acronym: ROBO-G
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: UZB-HLK: EVE-DJTT-002
Record Dates: First submitted 2022-09-19; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-04

CONDITIONS: Colorectal Surgery; Geriatric Assessment; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Older patients with colorectal cancer (Other): Patients undergo geriatric assessment including evaluation of cognitive function, functional status and quality of life
  Interventions: Diagnostic Test: Geriatric Assessment

INTERVENTIONS:
Diagnostic Test: Geriatric Assessment — Geriatric assessment to evaluate cognitive function, functional status and quality of life before and after surgery

SUMMARY:
The present study evaluates prospectively the impact of robotic surgery on functional outcome and quality of life in older patients that are operated for colorectal cancer;

ELIGIBILITY:
Inclusion Criteria:

* patients ≥ 70 years with colorectal cancer
* eligible for colorectal surgery after multidisciplinary board evaluation and patient consent

Exclusion Criteria:

* decline in cognitive function after geriatric evaluation
* emergency surgery
* life expectancy < 3 months

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in frailty status G8 status | Before and 3-6-12 months after surgery
  Measurement of functional status using the G8, Flemish version of the Triage Risk Screening Tool (fTRST)
Change in frailty status GFI status | Before and 3-6-12 months after surgery
  Measurement of functional status using the Groningen Frailty Indicator (GFI) Screening Tool (fTRST)
Change in Quality of Life | Before and 3-6-12 months after surgery
  Measurement of QoL using validated EORTC QoL questionnaire

SECONDARY OUTCOMES:
Percentage (%) of patients demonstrating functional improvement at 3, 6 and 12 months after surgery | 3-6-12 months after surgery
  Percentage (%) of patients demonstrating functional decline/improvement at 3, 6 and 12 months after surgery
Percentage of patients demonstrating functional recovery at 12 months after initial func-tional decline after surgery | 3-6-12 months after surgery
  Percentage of patients demonstrating functional recovery at 12 months after initial func-tional decline after surgery
Percentage of patients demonstrating a significant decrease/improvement of QoL at 3,6,12 months after surgery | 3-6-12 months after surgery
  Percentage of patients demonstrating a significant decrease/improvement of QoL at 3,6,12 months after surgery
Conversion-rate to open surgery | during surgery
  Number of patients where surgery can not be completed minimal invasive
Length of hospital stay | Immediate after surgery
  Time patient spends in hospital
Re-operation and re-admission rate | < 30 days after surgery
  need for re-intervention or hospitalisation after discharge
Evolution of post-operative cognition | 3, 6, 12 months post surgery
  Mini-cog clock test followed by Mini Mental State Evaluation (MMSE) if abnormal
Postoperative confusion rate | 7 days postoperative
  CAM-analysis
30- day post-operative morbidity (Clavien-Dindo classification) | < 30 days postoperative
  minor and major postoperative complications including anastomotic leakage
90- day post-operative mortality | < 90 days postoperative
  number of patients that die after surgery
1-year patient survival | 1 year postoperatively
  number of patients that are still alive one year after surgery
1-year disease free survival | 1 year postoperatively
  number of patients that do not show disease recurrence during the first postoperative year
Comparison in outcome parameters between frail patients (abnormal screening) versus fit patients | up till 12 months postoperatively
  Comparison in outcome parameters between frail patients (Groningen frailty indicator ≥ 4) versus fit patients (frailty indicator < 4)

OTHER OUTCOMES:
pathological analysis resection specimen | immediately after surgery
  tumor stage, lymph node yield, resection quality
blood loss | during surgery
  estimated blood loss during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Jacobs-Tulleneers-Thevissen, MD, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (2):
- Belgium (2):
  - Universitair Ziekenhuis Brussel, Brussels
  - Universitair Ziekenhuis Brussel, Jette

IPD SHARING:
Plan to Share IPD: No